CLINICAL TRIAL: NCT00487097
Title: Effect of EPA, GLA and Antioxidants on the Immune Response - Cellular and Molecular Mechanisms of Wound Healing in Critically Ill Patients.
Brief Title: The Effect of Antioxidants on the Immune Response and Wound Healing in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre singer, Professor, MD, Rabin Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4428
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Pressure Sores; Intensive Care
Keywords: intensive care; critically ill; fish oil; pressure sores
MeSH Terms: conditions — Pressure Ulcer; Critical Illness | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Enteral Nutrition with Omega 3 (Eicosapentanoic acid, docosahexaenoic acid)
  Interventions: Dietary Supplement: Eicosapentanoic acid, docosahexaenoic acid
- Control Group (No Intervention): Patients in control group will receive nutritional support composed of a standard formula

INTERVENTIONS:
Dietary Supplement: Eicosapentanoic acid, docosahexaenoic acid — Enteral nutrition formula enriched with Eicosapentanoic acid, docosahexaenoic acid
  Other Names: OXEPA
  Arms: Study Group

SUMMARY:
The purpose of this study is to investigate whether the addition of omega-3 and antioxidants to nutritional support in critically ill patients in the intensive care unit influences the immune and anti-inflammatory systems and so improves wound healing.

DETAILED DESCRIPTION:
A prospective randomized study to include 40 consecutive patients admitted to the general intensive care unit. The control group will receive nutritional support composed of a standard formula. The study group will receive nutritional support enriched with fish oil and anti-oxidants. The following variables will be assessed in all patients: demographics, severity of illness, assessment of bed sores. Blood tests will also be taken for the following: CD 8, CD 14, CD 18, CD 11a, CD49c, CD 49d. In addition, blood samples will be collected for TNF, IL-1b, IL-6, IL-8, and levels of C-reactive protein. Metabolic parameters such as resting energy expenditure, BMI, albumin, prealbumin, levels of zinc, relationship between omega 3 and omega 6. Theses test will be performed at time of ICU admission, days 7, 14 and 28 after admission.

The outcome: improved repair of pressure sores, together with improvement in objective parameters of immunity and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients in intensive care unit
* Grade 2 pressure sores

Exclusion Criteria:

* Immunosuppression with steroids or other agents
* Active bleeding
* Head trauma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Improvement of wound healing of pressure sores | within 28 days

SECONDARY OUTCOMES:
Improvement in parameters of immunity and inflammation | Within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Principal Investigator — Rabin Medical Center, Beilison Hospital, Israel
Locations (1):
- Rabin Medical center, Petah Tikva, Israel

REFERENCES:
- [Derived] Theilla M, Schwartz B, Cohen J, Shapiro H, Anbar R, Singer P. Impact of a nutritional formula enriched in fish oil and micronutrients on pressure ulcers in critical care patients. Am J Crit Care. 2012 Jul;21(4):e102-9. doi: 10.4037/ajcc2012187. PMID 22751375